CLINICAL TRIAL: NCT01246050
Title: Developing a Hub and Satellite Heart Failure Providers Network
Brief Title: "Hub and Satellite" Heart Failure Provider's Network Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RRP 09-170
Record Dates: First submitted 2010-11-19; First posted 2010-11-23 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Heart Failure
Keywords: Heart Failure; Outcome Assessment; Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Received HF Training (Experimental): Providers will receive 3 days of HF training, receive access to clinical pharmacist medication titration serviced and receive performance feedback
  Interventions: Other: HF training
- Arm 2: No HF Training (Active Comparator): CBOC Providers in the same CBOC who did not received HF Training, access to clinical pharmacist services or performance feedback
  Interventions: Other: No HF training

INTERVENTIONS:
Other: HF training — These are CBOC Providers who received HF Training as the active intervention. HF training includes didactic lectures, case discussions and interactive symposia, course materials including teaching material, textbooks, copies of HF clinical guidelines and patient education material for distribution, participation in HF Clinics and Inpatient Heart Failure Rounds. Providers were given access to clinical pharmacist services Including medication and disease teaching, adjustment and uptitration. There was quarterly analysis of patient compliance including individualized confidential, non-punitive feedback to providers from a set of prespecified core HF performance measures.
  Arms: Arm 1: Received HF Training
Other: No HF training — These are control providers drawn from the same CBOCs who have not received HF training, access to clinical pharmacist medication titration services or performance feedback
  Arms: Arm 2: No HF Training

SUMMARY:
The aim of this study is to serve as a pilot showing the feasibility of a "Hub and Satellite" Heart Failure (HF) Provider's Network which will aim to provide improved, evidence-based care to Veterans with HF. Primary Care Providers in the VA Community Based Outpatient Clinics (CBOCs) will undergo a brief period of intensive training in HF management and then practice in a network of primary care providers supported by the Regional HF Center.

DETAILED DESCRIPTION:
Background:

Congestive heart failure (HF) is a major public health problem. There is a pressing need to improve treatment of HF, but lifesaving therapies remain underused in clinical practice. The investigators proposed a novel, potentially cost-effective model of community-based, multidisciplinary, collaborative HF care - the "Hub and Satellite" Heart Failure Providers Network. Primary care providers trained in HF management would provide improved care to their clinic patients with HF in "satellite" clinics, supported by the Regional HF Center "hub".

Objectives:

1. To establish and demonstrate the feasibility of the "Hub and Satellite" Heart Failure Providers Network
2. To obtain data examining clinical effectiveness and barriers

Methods:

Volunteer community-based primary care providers underwent 3 days of HF management training at the regional HF center (Nashville), consisting of 21 hours of lectures, briefings, teaching sessions and case presentations. Multiple choice testing and a survey interview were completed at the beginning and end of training. Exclusive access was given to the services of a clinical pharmacist to titrate HF medications to clinical guideline-recommended doses.

Providers received updates on advances in HF management. A confidential feedback report on their performance was given to HF providers. Formative evaluation was performed through pre-educational and 4 subsequent telephone interviews with HF providers.

Decision Support System (DSS) data was used to identify patients with systolic HF (ejection fraction<40%) cared for by the HF providers; systolic HF patients in the same clinics cared for by non-HF trained providers were randomly selected as controls. Data on the care received over the one year period of follow-up was collected from DSS data and the computerized patient record system (CPRS).

Status:

One year of study follow-up has been completed. Primary data analysis is continuing. Work done to date has successfully demonstrated the feasibility of implementing a "Hub and Satellite" HF Providers network, including high provider satisfaction.

ELIGIBILITY:
Inclusion Criteria:

Healthcare providers (physicians, nurse practitioners, physician's assistants) who practice in a Community Based Outpatient Clinic (CBOC) in the Tennessee Valley Healthcare System, and are willing to undergo Heart Failure Training

Exclusion Criteria:

Community Based Outpatient Clinic (CBOC) Providers who are unable to attend the 3 day Heart Failure Training at the Regional Heart Failure Center.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry H Ooi, MD, Principal Investigator — VA Medical Center
Locations (1):
- Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Primary care providers practicing were recruited from Primary Care Clinics in the local VA healthcare system. Providers volunteered to be trained as Heart Failure providers and underwent specialized training in May 2010.
Groups:
- Arm 1: Received HF Training: CBOC Providers who have received HF Training
  3 days of training in HF management: HF training includes didactic lectures, case discussions and interactive symposia, course materials including teaching material, textbooks, copies of HF clinical guidelines and patient education material for distribution, participation in HF Clinics and Inpatient Heart Failure Rounds.
  Access to clinical pharmacist services: Including medication and disease teaching, adjustment and uptitration
  Quarterly analysis of physician compliance: Individualized confidential, non-punitive feedback to providers from a set of prespecified core HF performance measures.
- Arm 2: No HF Training: CBOC Providers in the same CBOC who have not received HF Training
Period: Overall Study
Arm/Group | Arm 1: Received HF Training | Arm 2: No HF Training
Started | 6 | 6 (Control providers were other providers in the same Primary Care Clinic, not enrolled in the study)
Completed | 6 | 6 (Control providers were other providers in the same Primary Care Clinic, not enrolled in the study)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Characteristics of Patients Followed by Providers in each Arm
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Received HF Training | Arm 2: No HF Training | Total
Number analyzed (Participants) | 129 | 129 | 258
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 65 [59 to 72] | 65 [62 to 74] | 65 [61 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 125 | 128 | 253
Coronary Artery Disease [Number; unit: participants]
  Coronary Artery Disease present | 101 | 97 | 198
  Coronary artery disease not present | 28 | 32 | 60
Hypertension [Number; unit: participants]
  Hypertension present | 119 | 119 | 238
  Hypertension not present | 10 | 10 | 20
Diabetes [Number; unit: participants]
  Diabetes present | 72 | 65 | 137
  Diabetes not present | 57 | 64 | 121
Median ejection fraction [Median (Inter-Quartile Range); unit: % left ventricular end-diastolic volume] | 30 [25 to 35] | 30 [25 to 35] | 30 [25 to 35]
Followed by Cardiology [Number; unit: participants]
  Number followed by Cardiology | 116 | 108 | 224
  Number not followed by Cardiology | 13 | 21 | 34
Followed by Advanced Heart Failure Clinic [Number; unit: participants]
  Followed by Heart failure Clinic | 26 | 37 | 63
  Not followed by Heart Failure Clinic | 103 | 92 | 195
HF Hospitalization past year [Number; unit: participants]
  No. with a HF hospitalization in the past year | 26 | 15 | 41
  No. without a HF hospitalization in the past year | 103 | 114 | 217

OUTCOME MEASURES:

1. Primary Outcome: Number of Superior Heart Failure Performance Outcome Quality Measures
Description: This was a pilot, qualitative study to assess the feasibility and preliminary outcomes of a program to train primary care providers in specialty care.
  9 Heart Failure Performance Outcome Quality Measures were studied:
  Patient weight measured at clinic visit; level of activity assessed; volume status assessed; Angiotensin Converting Enzyme Inhibitor/Angiotensin Receptor Blocker (ACEI/ARB) prescribed; ACEI/ARB at target dose; beta-blocker prescribed; beta-blocker at target dose; evidence-based beta-blocker used; coumadin prescribed in atrial fibrillation.
  Healthcare provider performance with each of the Performance Outcome Quality Measures was assessed at each study visit. Superior performance was defined as a higher score for each Measure on the follow-up visit compared to the baseline visit.
  The primary outcome of the study was considered to have been reached if 6 of the 9 outcome measures were superior to the baseline visit.
Time Frame: 12 months
Population: 129 patients cared for by HF trained primary care providers in Intervention Arm. 129 patients in the Control group, cared for by non-HF trained primary care providers.
Measure: Number; unit: number of outcome measures superior
Groups:
- Arm 1: Received HF Training: Patients followed by CBOC Providers who have received HF Training.
- Arm 2: No HF Training: Patients followed by CBOC Providers in the same CBOC who have not received HF Training
Arm/Group | Arm 1: Received HF Training | Arm 2: No HF Training
Number analyzed (Participants) | 129 | 129
number of outcome measures superior | 5 | 4

ADVERSE EVENTS:
Description: Neither providers or patients were monitored for adverse events
Arm/Group | Arm 1: Received HF Training | Arm 2: No HF Training
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
High performance on baseline metrics and infrequent primary care visits limited improvement opportunity.

Poor provider engagement and pharmacy service use may limit effect. High %Cardiology clinic co-management may limit study effectiveness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No